CLINICAL TRIAL: NCT00292994
Title: Exercise and Diet With Weight Loss in Metabolic Syndrome
Brief Title: Study of How Exercise or Weight Loss Effects Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yankton Clinical Research Alliance (Other)
Collaborators: University of South Dakota (Other); Yankton Medical Clinic (Other); Avera Sacred Heart Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 700-04-2001
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2006-02-16 (Estimated); Status verified 2006-01

CONDITIONS: Metabolic Syndrome; Insulin Resistance; Obesity
Keywords: Metabolic Syndrome; Hyperlipidemia; Type 2 diabetes mellitus; Insulin resistance; Weight loss; Obesity; Exercise; Hypertension
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Obesity; Hyperlipidemias; Diabetes Mellitus, Type 2; Weight Loss; Motor Activity; Hypertension | interventions — Exercise

INTERVENTIONS:
Behavioral: Exercise
Behavioral: Weight Loss

SUMMARY:
The Metabolic Syndrome (MS) is prevalent in the American population and is strongly associated with premature coronary disease. Lifestyle intervention, primarily exercise and dietary changes, are foundational treatment strategies for independent components of MS, but these interventions have not been thoroughly evaluated in MS. Even with very modest weight loss, in the setting of caloric restriction and exercise, marked improvement MS parameters have been noted. However, it is not known whether it is diet with weight loss or exercise that improves the metabolic derangements associated with MS. We propose a study designed to examine the relative impact of diet or exercise on the components of MS. Furthermore, it is known that psychological factors significantly impact the ability of patients to initiate and sustain lifestyle changes. We will monitor certain psychological states to evaluate their impact on the success of weight loss and sustainability of lifestyle changes throughout this study. Specific Aims: 1.) Evaluate the relative efficacy of diet with weight loss or exercise on improving the markers of metabolic syndrome. 2.) Determine of pre-existing psychological factors influence the effectiveness of diet with weight loss or exercise on the markers of metabolic syndrome. Design: Adult women (> 18 yrs) with a body-mass index (BMI)  30 kg/m2 will be assessed for MS and randomized to one of three groups (n = 34/group), Control (C), diet with weight loss alone (D), or exercise alone (E). The intervention groups will participate in supervised dietary changes designed for weight loss or exercise for 6 months. Anthropomorphic, serologic, and psychological parameters will be monitored and compared using ANOVA. Hypothesis: As indexed by the improvement in the laboratory markers of the components of metabolic syndrome, exercise alone has a more profound positive impact on Metabolic Syndrome then diet with weight loss alone.

DETAILED DESCRIPTION:
Research procedures: The interventions in this study will be caloric dietary restrictions intended to result in a 10% reduction of body weight within 6 months, or a supervised aerobic exercise program designed to improve cardiovascular fitness. The diet with weight loss group will meet with a registered dietician on a weekly basis for the first 2 months and then bi-weekly for the duration of the study for education and review of the subject's caloric intake. Similarly, the exercise group subjects will participate in weekly supervised aerobic exercise sessions. At these visits, a food logbook and an exercise logbook will be turned into the study staff to review. Prior to inclusion in the study, the patient's medical record will be reviewed for evidence of metabolic syndrome, specifically, recent lipid analysis, blood sugar, weight, height, waist circumference, and blood pressure. A self-report history and physical examination form, Perceived Behavior Control Scale, Self-Efficacy Scale, Beck Depression Inventory will also be included as part of the enrollment process and ongoing participation. Pre-intervention/initial screening includes fasting triglycerides, HDL, glucose, hs-CRP, Uric Acid, insulin, and plasma creatinine, 24-hour urine collection, blood pressure, waist and hip circumference, height, weight, VO2 max estimated from sub maximal standardized treadmill exercise test, Beck Depression Inventory, Perceived Behavioral Control Scale, Self-Efficacy Scale and Pre-intervention 3-day food record and physical activity questionnaire to assess baseline diet and activity levels. During study monitoring: daily exercise log (exercise group), assessed weekly, (determine the intensity, duration, and frequency of aerobic exercise), daily food log (diet with weight loss group), assessed for caloric intake, quarterly 3-day food records, assessed for caloric intake, and composition of fats, carbohydrates and proteins, quarterly blood pressure, weight, height, waist and hip circumference, quarterly fasting serum triglyceride, HDL, fasting serum glucose, and uric acid, and quarterly physical activity questionnaire, Beck Depression Inventory, Perceived Behavioral Control Scale, and Self-Efficacy Scale. Post-study assessment: fasting serum triglycerides, HDL, serum glucose, uric acid, hs-CRP, insulin, and plasma creatinine, 24-hour urine collection, body weight, height, and waist and hip circumference, VO2 max estimated from sub maximal standardized treadmill exercise test, and 3-day food record, physical activity questionnaire, Beck Depression Inventory, Perceived Behavioral Control Scale, and Self-Efficacy Scale. The control group will complete the pre and post measurements and the 3-day food record and physical activity questionnaire as required by the diet and exercise groups.

ELIGIBILITY:
Inclusion Criteria:Subjects who have been noted to meet the initial study criteria or have self-determined their eligibility from direct mailings, newspaper advertisement, or poster/flyers (female, age > 18, and a BMI of > 30) will contact the study coordinator. Subjects will come for an initial assessment where informed consent will be obtained. Their eligibility for inclusion or exclusion will be based on a determination that they do have metabolic syndrome and determined by the study coordinator (Janine Albers) and the principal investigators (Michael Hein or Jack Williams). This will be assessed by a review of their medical record, laboratory assessment, anthropomorphic measurements, and a focused History and Physical examination.

-

Exclusion Criteria: Cardiovascular: uncontrolled dyslipidemia (fasting triglycerides > 1000), type 1 diabetes, uncontrolled type 2 diabetes (Hgb A-1-c > 9.0%) or if on insulin, or uncontrolled hypertension (SBP > 180 or DBP > 100). Also, subjects with stable or unstable angina, a precedent myocardial infarction within six months of the study, or severe activity dyspnea, untreated major depression or patients with suicidal ideation, severe exercise-limiting inflammatory or degenerative arthritis, patients on anti-obesity medications or serotonin reuptake inhibitors, patients who are already involved in a regular aerobic exercise program (> 3 sessions of 30min/wk) or are involved with other weight loss programs with dietary regimen intervention as a component, e.g. Weight Watchers or other similarly structured weight loss programs. Pregnancy. Weigh greater than 350 pounds. -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2004-04; Study Completion 2006-01

PRIMARY OUTCOMES:
Metabolic Syndrome Score

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Hein, MD, Principal Investigator — Yankton Medical Clinic; John L Williams, PhD, Principal Investigator — Sanford School of Medicine at the University of South Dakota
Locations (1):
- Yankton Medical Clinic, Yankton, South Dakota, United States